CLINICAL TRIAL: NCT04304144
Title: CAEL101-203: A Phase 2, Open-label, Multicenter Dose Selection Study to Evaluate the Safety and Tolerability of CAEL-101 in Patients With AL Amyloidosis
Brief Title: A Study to Evaluate the Safety and Tolerability of CAEL-101 in Patients With AL Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAEL101-203
Record Dates: First submitted 2020-02-28; First posted 2020-03-11 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: AL Amyloidosis
Keywords: cyclophosphamide, bortezomib and dexamethasone (CyBorD); AL Amyloidosis; Amyloid, Light chain Amyloidosis; Mayo Stage IIIa; daratumumab; Mayo Stage II; Mayo Stage I
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Dexamethasone; daratumumab

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, sequential cohort, dose-selection study of CAEL-101 in Mayo Stage I, II and IIIa AL amyloidosis patients.
  The study is divided into two parts:
  * Part A defines the safety and tolerability of CAEL-101 in combination with SoC CyBorD and determines the RP3D
  * Part B evaluates the safety and tolerability of CAEL-101 in combination with SoC CyBorD and daratumumab
  Part A will employ a 3+3 dose escalation design. At least 3 patients will be enrolled in each dose cohort unless adverse events (AE) preventing further dosing are observed. Part B will enroll a minimum of 6 patients.
  Patients will be seen in the clinic weekly for 4 weeks to receive study drug infusions. Study drug infusions will be bi-weekly thereafter or every 4 weeks after 50 weeks, if participants switch to an alternative dosing schedule. Patients are treated until death, toxicity, symptomatic deterioration, Investigator, patient, or Sponsor decision to terminate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: CAEL-101 combined with SoC CyBorD (Experimental): CAEL-101 is administered as an intravenous (IV) infusion over approximately 2 hours. The initial cohort dose assignments of CAEL-101 will be: Cohort 1 - 500 mg/m^2 Cohort 2 - 750 mg/m^2 Cohort 3 - 1000 mg/m^2. CAEL-101 will be administered weekly for the first 4 weeks, and then every other week until end of study, in combination with the SoC CyBorD chemotherapy. Patients will be treated until death, unacceptable toxicity, symptomatic deterioration, Investigator decision, patient decision or Sponsor decision to terminate the study. Patients from Part A who are in the Continued Treatment Period and who, in the Investigator's judgment, should have their SoC treatment complemented with daratumumab may do so (Part B).
  Interventions: Drug: CAEL-101; Drug: SoC: cyclophosphamide, bortezomib, and Dexamethasone (CyBorD)
- Part B: CAEL-101 combined with SoC CyBorD and daratumumab (Experimental): CAEL-101 is administered as an intravenous (IV) infusion at the RP3D dose level. CAEL-101 will be administered weekly for the first 4 weeks, and then every other week until end of study, in combination with the SoC CyBorD chemotherapy and daratumumab. After completing approximately 50 weeks of treatment, participants may switch to an alternative maintenance dosing regimen of every four weeks (q4wk), if agreed upon by the Investigator and the Sponsor Medical Monitor. Patients will be treated until death, unacceptable toxicity, symptomatic deterioration, Investigator decision, patient decision or Sponsor decision to terminate the study.
  Interventions: Drug: CAEL-101; Drug: SoC: cyclophosphamide, bortezomib, and Dexamethasone (CyBorD); Drug: Daratumumab

INTERVENTIONS:
Drug: CAEL-101 — The investigational product, CAEL-101, is formulated as a sterile liquid solution of protein plus excipients for dilution in a single-use, stoppered, glass vial. Each 10 mL vial contains 300 mg of CAEL-101 at a concentration of 30 mg/mL. CAEL-101 will be diluted with commercially available 0.9% Normal Saline.
  Other Names: Anselamimab
Drug: SoC: cyclophosphamide, bortezomib, and Dexamethasone (CyBorD) — According to institutional standard of care.
Drug: Daratumumab — Treatment for AL amyloidosis
  Arms: Part B: CAEL-101 combined with SoC CyBorD and daratumumab

SUMMARY:
AL amyloidosis begins in the bone marrow where abnormal proteins misfold and create free light chains that cannot be broken down. These free light chains bind together to form amyloid fibrils that build up in the extracellular space of organs, affecting the kidneys, heart, liver, spleen, nervous system and digestive tract.

The primary purpose of this study is to determine the recommended dose of CAEL-101 to facilitate progression of further clinical trials and evaluate safety and tolerability of CAEL-101 in combination with the standard of care (SoC) cyclophosphamide-bortezomib-dexamethasone (CyBorD) chemotherapy and daratumumab .

DETAILED DESCRIPTION:
This is a multicenter, open-label, sequential cohort, dose-selection study of CAEL-101 in Mayo Stage I, Stage II and Stage IIIa AL amyloidosis patients. CAEL-101 will be administered in combination with the standard of care (SoC) cyclophosphamide-bortezomib-dexamethasone (CyBorD) chemotherapy and daratumumab.

The study is divided into two parts with the following objectives:

* Part A defines the safety and tolerability of CAEL-101 in combination with SoC CyBorD and determines the recommended Phase 3 dose (RP3D) of CAEL-101
* Part B evaluates the safety and tolerability of CAEL-101 in combination with SoC CyBorD and daratumumab

The study will also evaluate the pharmacokinetic profile of CAEL-101 and explore the PK profile of CAEL-101 when given bi-weekly (q2wk) versus once-monthly (q4wk) after the first 50 weeks.

Part A of the study will employ a 3+3 dose escalation design. At least 3 patients will be enrolled in each dose cohort unless adverse events (AE) preventing further dosing are observed. CAEL-101 will be administered in combination with the SoC CyBorD chemotherapy.

In Part B, a minimum of 6 new patients will receive CAEL-101 administered in combination with SoC CyBorD and daratumumab.

Patients from both Parts A and B will receive CAEL-101 therapy weekly and SoC throughout the safety observation period. CAEL-101 study drug infusions will continue, with dosing approximately every two weeks (q2wk) thereafter. SoC will continue per the Investigator's discretion. After completing approximately 50 weeks of treatment, participants may switch to an alternative maintenance dosing regimen of every four weeks (q4wk), if agreed upon by the Investigator and the Sponsor Medical Monitor.

Approximately 25 patients will be enrolled in the study at approximately 3 investigator sites.

Patients will be treated with CAEL-101 until death, unacceptable toxicity, symptomatic deterioration, Investigator decision, patient decision or Sponsor decision to terminate the study.

ELIGIBILITY:
Key Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study.

1. AL amyloidosis Mayo stage I, II or IIIa
2. For Part A only, measurable hematologic disease defined by at least one of the following:

   1. involved/uninvolved free light chain difference (dFLC) > 5mg/dL or
   2. free light chain (FLC) > 5mg/dL with abnormal Kappa/Lambda ratio or
   3. serum protein electrophoresis (SPEP) m- spike > 0.5 g/dL Patients with confirmed AL amyloid diagnosis without measurable disease may be enrolled with consultation and approval by the Sponsor Medical Monitor or their designee.
3. a. For Part A, currently on and continuing OR planned to start concurrent chemotherapy with CyBorD administered weekly as SoC. b. For Part B, currently on and continuing OR planned to start concurrent chemotherapy with CyBorD and daratumumab administered as SoC.

Key Exclusion Criteria:

Patients who meet any of the following criteria will not be permitted entry to the study.

1. Any form of secondary, hereditary, senile, localized, dialysis-related or leukocyte chemotactic factor 2-related (ALECT2) amyloidosis
2. Meets the International Myeloma Working Group (IMWG) definition of multiple myeloma. Patients with signs and/or symptoms attributable ONLY to amyloidosis and who do NOT meet IMWG definition of smoldering myeloma may be enrolled upon approval of the medical monitor.
3. Supine systolic blood pressure < 90 mmHg or symptomatic orthostatic hypotension, defined as a decrease in systolic blood pressure upon standing of > 20 mmHg despite medical management (e.g., midodrine, fludrocortisones) in the absence of volume depletion
4. Receiving dialysis
5. Myocardial infarction, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or percutaneous cardiac intervention with recent stent, coronary artery bypass grafting or major cerebrovascular accident within 6 months prior to screening
6. Left ventricular ejection fraction (LVEF) < 45 percent by echocardiogram or multigated acquisition scan (MUGA)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Stanford, California
  - Research Site, Detroit, Michigan
  - Research Site, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CAEL101-203&attachmentIdentifier=def51286-0693-4dce-8dd8-9043345d0b2e&fileName=CAEL101-203_Final_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: CAEL101 500 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 500 milligrams (mg)/square meter (m^2) administered weekly as an intravenous (IV) infusion the first 4 weeks (dose limiting toxicity [DLT] observation period), and thereafter received CAEL-101 at the recommended phase 3 dose (RP3D) (1000 mg/m^2) every other week until the end of study, in combination with the standard of care (SoC) CyBorD (cyclophosphamide, bortezomib, dexamethasone) chemotherapy.
- Part A: CAEL101 750 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 750 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period), and thereafter received CAEL-101 at the RP3D (1000 mg/m^2) every other week until the end of study, in combination with the SoC CyBorD chemotherapy.
- Part A: CAEL101 1000 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 1000 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period), and then every other week until the end of study, in combination with the SoC CyBorD chemotherapy.
- Part B: CAEL-101 Combined With SoC CyBorD and Daratumumab: Participants received CAEL-101 at the RP3D (1000 mg/m^2) administered weekly as an IV infusion for the first 4 weeks, and then every other week until end of study, in combination with the SoC CyBorD chemotherapy and daratumumab.
Period: DLT Observation Period
Arm/Group | Part A: CAEL101 500 mg/m^2 Combined With SoC CyBorD | Part A: CAEL101 750 mg/m^2 Combined With SoC CyBorD | Part A: CAEL101 1000 mg/m^2 Combined With SoC CyBorD | Part B: CAEL-101 Combined With SoC CyBorD and Daratumumab
Started | 4 | 3 | 6 | 0
Received At Least 1 Dose of Study Drug | 4 | 3 | 6 | 0
Completed (Study Completion) | 4 | 2 | 6 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Continued Treatment Period
Arm/Group | Part A: CAEL101 500 mg/m^2 Combined With SoC CyBorD | Part A: CAEL101 750 mg/m^2 Combined With SoC CyBorD | Part A: CAEL101 1000 mg/m^2 Combined With SoC CyBorD | Part B: CAEL-101 Combined With SoC CyBorD and Daratumumab
Started | 4 | 2 | 6 | 12
Completed | 1 | 1 | 4 | 6
Not Completed | 3 | 1 | 2 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 3
Not completed — Other than specified | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were treated with at least 1 dose of CAEL-101.
Groups:
- Part A: CAEL101 500 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 500 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period), and thereafter received CAEL-101 at the RP3D (1000 mg/m^2) every other week until the end of study, in combination with the SoC CyBorD.
- Part A: CAEL101 1000 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 1000 mg/m^2 administered weekly as an IV infusion the first 4 weeks, and then every other week until the end of study, in combination with the SoC CyBorD chemotherapy.
- Total: Total of all reporting groups
Arm/Group | Part A: CAEL101 500 mg/m^2 Combined With SoC CyBorD | Part A: CAEL101 750 mg/m^2 Combined With SoC CyBorD | Part A: CAEL101 1000 mg/m^2 Combined With SoC CyBorD | Part B: CAEL-101 Combined With SoC CyBorD and Daratumumab | Total
Number analyzed (Participants) | 4 | 3 | 6 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 1 | 8 | 14
  >=65 years | 0 | 2 | 5 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 4 | 7
  Male | 4 | 2 | 4 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 6 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 3 | 2 | 6 | 12 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) and Adverse Events (AEs), and AEs Leading to Treatment Discontinuation
Description: An adverse event (AE) was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), or an important medical event or reaction. A TEAE was defined as an AE that started after the first dose of treatment and before the last dose of study drug +140 days. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: First dose of study drug until 140 days after last dose of study drug (Maximum exposure: 38.90 months for Part A and 32.50 months for Part B)
Population: Safety Set included all participants who were treated with at least 1 dose of CAEL-101. AE data were collected for the participants in the DLT period (Part A) by dose separately. Additionally, the AE data for participants in the DLT period were also collected regardless of dose level received along with the AE data collected during the Part A Continued Treatment (Part A) period as an Overall arm.
Measure: Count of Participants; unit: Participants
Groups:
- DLT Period (Part A): CAEL-101 500 mg/m^2: Participants received CAEL-101 500 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period).
- DLT Period (Part A): CAEL-101 750 mg/m^2: Participants received CAEL-101 750 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period).
- DLT Period (Part A): CAEL-101 1000 mg/m^2: Participants received CAEL-101 1000 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period).
- Overall (Part A): DLT + Continued Treatment Period: CAEL-101 Combined With SoC CyBorD: Participants received CAEL-101 during the DLT period weekly as an IV infusion the first 4 weeks, and thereafter received CAEL-101 at the RP3D (1000 mg/m^2) every other week until the end of study, in combination with the SoC CyBorD (cyclophosphamide, bortezomib, dexamethasone) chemotherapy.
- Continued Treatment Period (Part B): CAEL-101 Combined With SoC CyBorD and Daratumumab: Participants received CAEL-101 at the RP3D (1000 mg/m^2) administered weekly as an IV infusion for the first 4 weeks, and then every other week until end of study, in combination with the SoC CyBorD chemotherapy and daratumumab.
Arm/Group | DLT Period (Part A): CAEL-101 500 mg/m^2 | DLT Period (Part A): CAEL-101 750 mg/m^2 | DLT Period (Part A): CAEL-101 1000 mg/m^2 | Overall (Part A): DLT + Continued Treatment Period: CAEL-101 Combined With SoC CyBorD | Continued Treatment Period (Part B): CAEL-101 Combined With SoC CyBorD and Daratumumab
Number analyzed (Participants) | 4 | 3 | 6 | 13 | 12
Participants
  Any TEAEs | 4 | 3 | 6 | 13 | 12
  Treatment-emergent SAEs | 0 | 0 | 2 | 9 | 7
  AEs Leading to Treatment Discontinuation | 0 | 0 | 0 | 3 | 1

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT) During the First 4 Weeks of Therapy
Description: A DLT was defined as any Grade 3 or greater study intervention-related AE that was clinically significant.
Time Frame: 4 weeks
Population: Safety Set included all participants who were treated with at least 1 dose of CAEL-101.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: CAEL-101 500 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 500 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period), and thereafter received CAEL-101 at the RP3D (1000 mg/m^2) every other week until the end of study, in combination with the SoC CyBorD.
- Part A: CAEL-101 750 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 750 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period), and thereafter received CAEL-101 at the RP3D (1000 mg/m^2) every other week until the end of study, in combination with the SoC CyBorD chemotherapy.
- Part A: CAEL-101 1000 mg/m^2 Combined With SoC CyBorD: Participants received CAEL-101 1000 mg/m^2 administered weekly as an IV infusion the first 4 weeks, and then every other week until the end of study, in combination with the SoC CyBorD chemotherapy.
Arm/Group | Part A: CAEL-101 500 mg/m^2 Combined With SoC CyBorD | Part A: CAEL-101 750 mg/m^2 Combined With SoC CyBorD | Part A: CAEL-101 1000 mg/m^2 Combined With SoC CyBorD | Part B: CAEL-101 Combined With SoC CyBorD and Daratumumab
Number analyzed (Participants) | 4 | 3 | 6 | 12
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of CAEL-101
Time Frame: Predose through Week 1 and through Week 20
Population: The Pharmacokinetic Set (PKS) included all participants who had at least 1 measurable plasma concentration. Number analyzed = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms (µg)/milliliter (mL)
Groups:
- Part A: CAEL-101 500 mg/m^2: Participants received CAEL-101 500 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period), and thereafter received CAEL-101 at the RP3D (1000 mg/m^2) every other week until the end of study.
- Part A: CAEL-101 750 mg/m^2: Participants received CAEL-101 750 mg/m^2 administered weekly as an IV infusion the first 4 weeks (DLT observation period), and thereafter received CAEL-101 at the RP3D (1000 mg/m^2) every other week until the end of study.
- Part A: CAEL-101 1000 mg/m^2: Participants received CAEL-101 1000 mg/m^2 administered weekly as an IV infusion the first 4 weeks, and then every other week until the end of study.
- Part B: CAEL-101 1000 mg/m^2: Participants received CAEL-101 at the RP3D (1000 mg/m^2) administered weekly as an IV infusion for the first 4 weeks, and then every other week until end of study.
Arm/Group | Part A: CAEL-101 500 mg/m^2 | Part A: CAEL-101 750 mg/m^2 | Part A: CAEL-101 1000 mg/m^2 | Part B: CAEL-101 1000 mg/m^2
Number analyzed (Participants) | 4 | 3 | 6 | 12
micrograms (µg)/milliliter (mL)
  Week 1 | 126 (16.7) | 255 (136) | 244 (92.8) | 280 (63.0)
  Week 20: number analyzed (Participants) | 0 | 0 | 6 | 9
  Week 20 |  |  | 580 (270) | 552 (194)

4. Secondary Outcome: Area Under Plasma Concentration-time Curve Over Dosing Interval (AUCtau) of CAEL-101
Time Frame: Predose through Week 1 and through Week 20
Population: The PKS included all participants who had at least 1 measurable plasma concentration. Number analyzed = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: hours*µg/mL
Arm/Group | Part A: CAEL-101 500 mg/m^2 | Part A: CAEL-101 750 mg/m^2 | Part A: CAEL-101 1000 mg/m^2 | Part B: CAEL-101 1000 mg/m^2
Number analyzed (Participants) | 4 | 3 | 6 | 12
hours*µg/mL
  Week 1 | 14400 (1290) | 27600 (12800) | 28600 (12700) | 29400 (6640)
  Week 20: number analyzed (Participants) | 0 | 0 | 6 | 9
  Week 20 |  |  | 147000 (69600) | 139000 (66700)

ADVERSE EVENTS:
Time Frame: First dose of study drug until 140 days after last dose of study drug (Maximum exposure: 38.90 months for Part A and 32.50 months for Part B)
Description: Safety Set included all participants who were treated with at least 1 dose of CAEL-101. AE data were collected for the participants in the DLT period (Part A) by dose separately. Additionally, the AE data for participants in the DLT period were also collected regardless of dose level received along with the AE data collected during the Part A Continued Treatment (Part A) period as an Overall arm.
Arm/Group | DLT Period (Part A): CAEL-101 500 mg/m^2 | DLT Period (Part A): CAEL-101 750 mg/m^2 | DLT Period (Part A): CAEL-101 1000 mg/m^2 | Overall (Part A): DLT + Continued Treatment Period: CAEL-101 Combined With SoC CyBorD | Continued Treatment Period (Part B): CAEL-101 Combined With SoC CyBorD and Daratumumab
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/6 | 1/13 | 2/12
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 1/6 | 9/13 | 7/12
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 6/6 | 13/13 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLT Period (Part A): CAEL-101 500 mg/m^2 (N=4) | DLT Period (Part A): CAEL-101 750 mg/m^2 (N=3) | DLT Period (Part A): CAEL-101 1000 mg/m^2 (N=6) | Overall (Part A): DLT + Continued Treatment Period: CAEL-101 Combined With SoC CyBorD (N=13) | Continued Treatment Period (Part B): CAEL-101 Combined With SoC CyBorD and Daratumumab (N=12)
Splenic Haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 3 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Nodal Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Catheter Site Haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Testicular abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin T Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Depressed Level of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Clostridium Difficile Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLT Period (Part A): CAEL-101 500 mg/m^2 (N=4) | DLT Period (Part A): CAEL-101 750 mg/m^2 (N=3) | DLT Period (Part A): CAEL-101 1000 mg/m^2 (N=6) | Overall (Part A): DLT + Continued Treatment Period: CAEL-101 Combined With SoC CyBorD (N=13) | Continued Treatment Period (Part B): CAEL-101 Combined With SoC CyBorD and Daratumumab (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 7 (11) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Ear Haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 (2) | 0 (0)
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 3 (4) | 3 (4)
Cataract (Eye disorders) | 0 | 1 | 0 | 1 (1) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Vitreous Floaters (Eye disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 7 (11) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 8 (18) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 7 (11) | 4 (7)
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 5 (5) | 2 (3)
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (3)
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (3) | 0 (0)
Fatigue (General disorders) | 1 | 0 | 1 | 8 (12) | 5 (7)
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 3 (6) | 5 (9)
Localised Oedema (General disorders) | 0 | 0 | 1 | 2 (3) | 0 (0)
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 4 (5) | 2 (2)
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3 (5) | 3 (8)
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 3 (12) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 3 (3) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 (13) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (3) | 3 (5)
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 (2) | 2 (2)
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 | 0 | 1 | 7 (10) | 1 (1)
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 3 (6) | 4 (10)
Weight Decreased (Investigations) | 0 | 0 | 0 | 2 (2) | 3 (4)
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 3 (3) | 1 (1)
Weight Increased (Investigations) | 0 | 0 | 0 | 3 (4) | 1 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1 | 2 (2) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 (0) | 2 (2)
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 1 | 1 (1) | 1 (1)
Neutrophil Count Increased (Investigations) | 0 | 0 | 0 | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 (7) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 (5) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 (10) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 (5) | 3 (3)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 (2) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 4 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 (2) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 2 (5)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (2) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 2 (2)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 6 (6) | 3 (4)
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 4 (4) | 3 (4)
Headache (Nervous system disorders) | 1 | 1 | 0 | 3 (3) | 3 (5)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 (2) | 2 (3)
Disturbance In Attention (Nervous system disorders) | 0 | 0 | 0 | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 2 (4)
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 5 (5) | 2 (3)
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 7 (12) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 6 (10) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 (5) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (2) | 2 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 (7) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 2 (3)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (2) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 5 (8) | 2 (2)
Hypertension (Vascular disorders) | 0 | 1 | 0 | 3 (6) | 2 (4)
Haematoma (Vascular disorders) | 0 | 0 | 0 | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Pulmonary Edema (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0
Hemoptysis (General disorders) | 0 | 1 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Muscle Cramp (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Peripheral Neuropathy NOS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT04304144/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT04304144/SAP_001.pdf